CLINICAL TRIAL: NCT04144816
Title: Exploring the Role of Socio Demographic, Clinical Risk Factors, Cord Specific Antibody at Birth, and Virus Characteristic, in Respiratory Syncytial Virus (RSV) in Hospitalized vs Ambulant Infants
Brief Title: Predictors of Respiratory Syncytial Virus (RSV) Hospitalizations in Infants
Acronym: PRSVH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PRSVH_2019
Record Dates: First submitted 2019-10-18; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Syncytial Virus Respiratory Infection; RSV Infection; Respiratory Syncytial Virus Infections; RSV Bronchiolitis
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Cordon (remained after diagnosis use) Respiratory samples (remained after diagnosis use)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Passive Birth Cohort: This will be a multicenter, prospective, observational cohort study conducted across the Lyon Public hospital maternity (HFME : Hospital for women, mother and children, Croix-Rousse, Lyon-Sud) recruited from the general population.
  Infants born between October 2019 and march 2020. At birth the remains (after diagnosis use) of cord blood samples will be store. Groups of RSVh cases and control will be class at one year of age using the hospital data (RSV must be confirmed by RT-PCR). Parents will be informed of the protocol. If enrolled available hospital data will be use and RSV serology testing perform on the store blood cordon.
  Interventions: Other: Not applicable (no intervention)

INTERVENTIONS:
Other: Not applicable (no intervention) — Not applicable (no intervention)

SUMMARY:
The VRS (Respiratory Syncytial Virus) study group in Lyon is a working that aims to understand, predict and prevent the burden of disease caused by human respiratory syncytial virus (RSV) infection in infants. Incidence of RSV-associated hospitalization in the first year of life was estimated at 14.5 (95% CI 13.4-15.6) per 1000 births in a cohort study in Lyon, France. Related direct medical annual costs were estimated for this cohort at 364,269€, mostly attributed to children born during the RSV season (231,959€) and children born premature (108,673€). This study will combine existing hospital specimens and databases to determine the respective role of socio demographic factors, clinical risk factors, level of cord specific antibody at birth, and virus characteristic in the Respiratory Syncytial Virus (RSV) Hospitalization outcome in Infants.

Regarding the introduction of a new RSV vaccine and RSV-specific neutralizing antibodies, these data are of prime importance to guide future vaccine policies.

DETAILED DESCRIPTION:
Objective:

To determine the main predictors of Respiratory Syncytial Virus (RSV) Hospitalizations in Infants

Study design:

Prospective epidemiological, observational, one-center cohort study with sample collection.

Study population:

Birth cohort of infants born in Lyon before and during the RSV circulation period (October to march) with a follow-up until one year old (from birth until the age of 1 year maximum):

* Estimate Birth cohort (n=5,000).
* Estimate number of RSVH case (n=110).
* Estimate number of Blood cordon associated with a RSVH (Respiratory Syncytial Virus Human) case (n=60)

ELIGIBILITY:
Inclusion Criteria:

* Children born alive at participating centers.
* Parents living in the Rhone Alpes Auvergne region

Exclusion Criteria:

* Parents non-willing to participate
* Parents living outside the region

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Birth cohort of 5 000 infants of the general population recruited from the HCL (Public hospital of Lyon) maternity wards during the first days after birth
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Number of cases included in the cohort with RT-PCR (Retrotranscription) confirmed RSV hospitalization occurring from birth until the age of 1 year | 1 year after inclusion
  Cases were defined as a new admission to one of the conventional pediatric hospital departments with a RSV positive sample during the hospital stay the first 3 years of life.
Number of cases included in the cohort with RT-PCR confirmed RSV hospitalization occurring from birth until the age of 3 years. | 3 years after inclusion
  Cases were defined as a new admission to one of the conventional pediatric hospital departments with a RSV positive sample during the hospital stay the first 3 years of life.

SECONDARY OUTCOMES:
Quantitative level of anti-RSV IgG measure | 3 years after inclusion
  The quantitative level of anti-RSV IgG at birth in blood cord cordon will be compare between the cases group and the control group (No admission to one of the conventional pediatric hospital departments with a RSV positive sample during the hospital stay the first 3 years of life)
Quantitative level of anti-RSV IgG (Immunoglobulin G) measure | 3 years after inclusion
  The quantitative level of anti-RSV IgG at birth in blood cord cordon will be compare between the cases group and the control group (No admission to one of the conventional pediatric hospital departments with a RSV positive sample during the hospital stay the first 3 years of life)